CLINICAL TRIAL: NCT04426734
Title: Evaluation of DEXTENZA on the Management of Pain and Inflammation in Patients With Anterior Uveitis Compared to Standard of Care Topical Corticosteroids
Brief Title: Evaluation of DEXTENZA in the Management of Pain and Inflammation in Patients With Anterior Uveitis Compared to Standard of Care Topical Corticosteroids
Acronym: DiverT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: New England Retina Associates (Other)
Collaborators: Ocular Therapeutix (Unknown)
Responsible Party: Principal Investigator, John Huang, MD, Ophthalmologist and Clinical Associate Professor, New England Retina Associates
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OT V1
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Non-infectious Anterior Uveitis

STUDY DESIGN:
Intervention Model Description: Sustained Release Dexamethasone, 0.4 mg, intracanalicular insert
  Thirty patients with anterior uveitis will be randomized to receive either:
  Sustained Released 0.4 mg Dexamethasone intracanalicular insert in both upper and lower punctum.
  OR
  Topical corticosteroid (Pred Forte, prednisolone acetate 1%) standard of care tapered treatment regimen of
  8x/day week 1 4x/day week 2 2x/day week 3
  1x/day week 4
  Visit schedule: Baseline, Day 3, Day 7, Day 14, and Day 30
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Dextenza (Experimental): Sustained Released 0.4 mg Dexamethasone intracanalicular insert in both upper and lower punctum.
  Visit schedule: Baseline, Day 3, Day 7, Day 14, and Day 30
  Interventions: Device: Dextenza Dexamethasone Implant
- Topical Pred Forte 1% (Active Comparator): Topical corticosteroid (Pred Forte, prednisolone acetate 1%) standard of care tapered treatment regimen of
  8x/day week 1 4x/day week 2 2x/day week 3
  1x/day week 4
  Visit schedule: Baseline, Day 3, Day 7, Day 14, and Day 30
  Interventions: Drug: Topical Prednisolone Acetate 1%

INTERVENTIONS:
Device: Dextenza Dexamethasone Implant — The area of the punctum is first anesthetized with eye drops. A localized injection of lidocaine in perform once the surface of the punctum is numbed with the eyedrop. After 5-10 minutes, the corner of the eyelid and the region of the punctum will be fully anesthetic. The upper and lower punctum are then dilated with a punctum dilator to facilitate the insertion of the DEXTENZA medication. The DEXTENZA medication is then inserted using smooth forceps into the dilated opening of the upper and lower punctum. Once the DEXTENZA is inserted into the both the upper and lower punctum, the procedure is down. No repeated insertion of the DEXTENZA is required for the study.
  Arms: Dextenza
Drug: Topical Prednisolone Acetate 1% — Topical corticosteroid (Pred Forte, prednisolone acetate 1%) standard of care tapered treatment regimen of
  8x/day week 1 4x/day week 2 2x/day week 3
  1x/day week 4
  Visit schedule: Baseline, Day 3, Day 7, Day 14, and Day 30
  Other Names: Topical Pred Forte 1%
  Arms: Topical Pred Forte 1%

SUMMARY:
This a prospective study review of the clinical efficacy of DEXTENZA for the treatment of anterior uveitis compared to the standard of care topical corticosteroid treatment

DETAILED DESCRIPTION:
Patients with anterior uveitis are typically treated aggressively with every 1-2 hour (while the patient is awake) potent topical steroid agents, during initial stage of inflammation, and evaluated at frequent intervals, with a schedule of steroid tapering dictated by clinical response. The most common topical corticosteroid prescribed for the treatment of anterior uveitis are prednisolone acetate 1%, dexamethasone 0.1%, prednisolone sodium phosphate 1% and Difluprednate 0.05%. However, topical treatments are limited by the potential for patient non-adherence and variation in drug concentrations due to the intermittent or suspension of use nature of application. A corticosteroid insert placed in the inferior and superior canaliculi provides the advantages of reliable and continuous drug delivery for 24 hours a day for 30 days without the need for patients to adhere to a treatment regimen. Dextenza is a sustained-release dexamethasone intracanalicular insert recently approved by the FDA for pain and inflammation post ophthalmic surgery. Dextenza was shown to decrease inflammation and pain compared with placebo following cataract surgery in a multicenter randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Active non-infectious anterior uveitis
* Able to provide signed written consent prior to participation in any study-related procedures.

Exclusion Criteria:

* Have active intermediate, posterior uveitis, or panuveitis
* Have infectious anterior uveitis
* Have used topical corticosteroid treatment up to 48 hours prior to the baseline visit
* Have used oral corticosteroid within the past 14 days prior to baseline visit (Patients using stable doses of inhaled corticosteroids for 30 days prior to baseline visit can be included in the study)
* Have received intravitreal or sub-Tenon corticosteroid treatment prior to baseline visit or Ozurdex ® in the study eye within the 6 months prior to the baseline visit
* Are currently using prescribed nonsteroidal anti-inflammatory agents or prescribed immunosuppressive agents, unless the dose has been stable for the last 6 weeks and no change in dosing is anticipated for the duration of the study
* Have severe/serious ocular pathology or medical condition which may preclude study completion
* Dacriocystitis
* Are pregnant or lactating female, or female of childbearing age using inadequate birth control method
* Have participated in another investigational device or drug study within 30 days of the baseline visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Response of Anterior Uveitis to Treatment | 30 days
  Proportion of Subjects with Anterior Chamber Cell Grade of 0 from baseline at days 3, 7, 14, and 30

SECONDARY OUTCOMES:
Improve 2 grade levels by SUN grading system | 30 days
  • Proportion of subjects with a reduction in anterior chamber cell count score of 2 or more SUN grading scale levels from baseline at Days 3, 7, 14, and 30
Mean change in cells | 30 days
  Mean change from baseline in anterior chamber cell scores at days 3, 7, 14 and 30.
Mean change in flare | 30 days
  Mean change from baseline in anterior chamber cell flare scores at days 3, 7, 14 and 30.
Time to zero inflammation | 30 days
  Time to anterior cell count score of zero from baseline over time
OCT | 30 days
  Mean change from baseline in retinal thickness as measured by Optical Coherence Tomography (OCT)
CME | 30 days
  Proportion of patients who develop cystoid macular edema from baseline at days 3, 7, 14, and 30
Proportion of resolution of CME | 30 days
  Proportion of patients with resolution of retinal thickness (normalized retinal thickness) from baseline through day 30 as measured by OCT
Mean change in Visual Acuity | 30 days
  Mean change in BCVA from baseline at days 3, 7, 14 and 30.
IOP | 30 days
  Mean change in IOP from baseline at days 3, 7, 14 and 30.
NEI-VQ-25 | 30 days
  Mean change in NEI-VFQ 25 from baseline to day 30
Rescue therapy | 30 days
  Percentage of study eyes requiring rescue treatment from baseline through day 30
Adverse events | 30 days
  Incidence and severity of adverse events

IPD SHARING:
Plan to Share IPD: No
This data will be analyzed and published by the principle investigator.